CLINICAL TRIAL: NCT00464529
Title: Peri-Operative Accuracy and Safety of Real Time Continuous Glucose Monitoring System in Cardiac Surgical Patients. A Pilot Study
Brief Title: Accuracy and Safety of Real Time Continuous Glucose Monitoring Before, During and After Surgery
Acronym: GluContinu
Status: Completed | Type: Observational
Sponsor: Medical Research Foundation, The Netherlands (Other)
Collaborators: Medtronic (Industry)
Other Study IDs: 06.0741
Record Dates: First submitted 2007-04-20; First posted 2007-04-23 (Estimated); Last update posted 2007-11-07 (Estimated); Status verified 2007-05

CONDITIONS: Glucose Metabolism Disorders; Perioperative Care
Keywords: blood glucose; hyperglycemia; hypoglycemia; Perioperative care; inpatient
MeSH Terms: conditions — Glucose Metabolism Disorders; Hyperglycemia; Hypoglycemia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Real-Time Continuous Glucose monitoring System (RT-CGMS)

SUMMARY:
The purpose of this study is to determine the safety and accuracy of the Real-Time Continuous Glucose monitoring System (RT-CGMS)in measuring glucose in patients scheduled for surgery; before, during and after surgery.

DETAILED DESCRIPTION:
Rationale:Strict glycaemic control improves outcome of critically ill patients. Real Time Continuous Glucose monitoring System (RT-CGMS) is a novel system which can provide health care professionals with real time information about the blood glucose level without the need for multiple invasive measurements. Furthermore, with continuous monitoring it is possible to identify trends in glycaemic profiles. Its accuracy and safety have never been tested in a population of patients admitted to an intensive care unit.

Objective:To investigate the accuracy and safety of the RT-CGMS in patients scheduled for elective cardiac surgery. Our secondary objective is to define the possible factors interfering with reliable and adequate glucose measurements and to investigate the effect of RT-CGMS on glucose control.

Study design: Open label, randomised controlled trial. Study population:Patients scheduled for elective cardiac surgery. Intervention:After informed consent and randomisation, all patients will have the RT-CGMS inserted pre-operatively. In one group (Control group; 15 subjects), the RT-CGMS will be blinded, so that no information on blood glucose values measured and stored by the RT-CGMS will be available to care-givers, investigators or patients during the study period. In the other group (Active group, 15 subjects), the RT-CGMS will not be blinded. The system will alert whenever a glucose level falls below or rises above preset values. Sensor values are not intended to be used directly for making therapy adjustments. Whenever a value is below or above the preset value, the blood glucose level will be measured using separate blood analysis and therapy adjustments based on this value will be done according to the (ICU) protocol.

Study endpoints: Correlation between data obtained with the RT-CGMS and the conventional method. Degree of glucose control defined as the time spent in normoglycaemia, hypoglycaemia and hyperglycaemia, as recorded both with sensor measurements and ward measurements. Occurrence of significant clinical events and its effect on RT-CGMS.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective cardiac surgery
* Age >18 years
* Both patients with diabetes mellitus as non-diabetic patients are eligible

Exclusion Criteria:

* Failure to obtain informed consent
* pre-admission insulin treatment for diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-05; Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henk J Bilo, MD PhD, FRCP, Principal Investigator — Isala Clinics, Diabetes Centre
Locations (1):
- Isala Clinics, Weezenlanden location, Zwolle, Netherlands